CLINICAL TRIAL: NCT07303361
Title: Effects of Active Techniques and Mandibular and Cervical Motor Control on Pain, Functionality, and Associated Psychosocial Factors in Patients With Temporomandibular Disorder and Bruxism. Randomized Controlled Clinical Trial
Brief Title: Effect of Active Mandibular Techniques and Specific Cranio-cervical Therapeutic Exercise in Patients With Temporomandibular Disorders and Bruxism (AMaCe-TB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Gerencia Regional de Salud de Castilla y Leon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMaCe-TB
Record Dates: First submitted 2025-12-02; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Disorder (TMD)
Keywords: temporomandibular disorder; bruxism; pain control
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific technique Group (Experimental): Patients will undergo the mandibular muscle energy technique, as well as specific craniocervical motor control exercises.
  Interventions: Procedure: Mandibular Muscle Energy Technique
- Stardard clinical treated group (Placebo Comparator): Patients will receive standard clinical treatment and, in addition, a single session of treatment using a modified suboccipital inhibition technique plus non-specific cervical mobility exercises at home (flexion, extension, and rotation) for 4 weeks.
  Interventions: Procedure: Modified suboccipital inhibition technique

INTERVENTIONS:
Procedure: Mandibular Muscle Energy Technique — The mandibular muscle energy technique lasts approximately 3-4 minutes. The physical therapist stands next to the patient to use the jaw motion rehabilitation system, which will allow the technique to be applied through a system of controlled opening and resistance to closure, with a real assessment of the balance of mouth opening. The patient will be asked to open their mouth and it will be gently increased, while the patient's forehead is fixed, up to the patient's joint opening range. From this position, the patient will be asked to perform an isometric contraction of the masticatory muscles for approximately 3-5 seconds. This procedure will be performed in three cycles, with three contractions per cycle and a rest period between contractions of approximately 3-5 seconds. Patients will perform specific craniocervical motor control exercises for 4 weeks and will be monitored during weekly visits, where manual treatment will be performed using the mandibular muscle energy technique.
  Arms: Specific technique Group
Procedure: Modified suboccipital inhibition technique — The modified suboccipital inhibition technique will be performed at the beginning as a placebo technique. This technique will last 5 minutes. For this technique, the patient will lie on the table. The aim of this technique is to provide a stimulus as similar as possible to the original suboccipital inhibition technique, but without the force of movement. The patient will keep their eyes closed for the duration of the technique.
  Arms: Stardard clinical treated group

SUMMARY:
Temporomandibular Disorders (TMD) are a common source of pain and functional limitation affecting the stomatognathic system. They frequently lead to difficulties in mastication, decreased quality of sleep, limited mandibular mobility, and restrictions in daily activities. These symptoms are often aggravated in patients with associated bruxism. Chronic involvement of the temporomandibular joint and surrounding structures can also negatively influence cervical posture and motor control due to the neurophysiological connections between the cranio-cervical region and mandibular biomechanics. This study is designed to evaluate whether active mandibular techniques, specifically the Muscle Energy Technique (MET) applied with the support of the jaw motion rehabilitation system, combined with a cranio-cervical therapeutic exercise program, may improve pain, function, and motor behavior in patients with chronic TMD and bruxism.

The trial will be conducted as a randomized controlled study with two parallel groups. The experimental group will receive a mandibular MET intervention delivered once weekly for four weeks, using an active resistance and controlled movement protocol based on three cycles of isometric contraction and passive stretching. In addition, participants will perform daily cranio-cervical motor control exercises at home, with weekly supervision. These exercises aim to enhance neuromuscular regulation of deep cervical flexors and extensors and improve cervical dissociation, symmetry, and alignment. The control group will receive standard clinical care supplemented by a single session of a modified suboccipital inhibition technique acting as a placebo procedure. They will also perform non-specific cervical mobility exercises at home over a four-week period.

The primary outcome will be the change in Pressure Pain Threshold (PPT) measured with a pressure algometer at trigger points located in the trapezius, masseter, external pterygoid, and digastric muscles. Secondary outcomes will include maximum mouth opening, pain intensity using a visual analog or numeric rating scale, craniocervical postural control assessed through standardized motor control evaluations, and mandibular movement behavior analyzed through visual or device-assisted kinematic assessment. Measurements will be taken at baseline, immediately after the intervention period, and during a follow-up assessment.

Participants will be adults aged 18 to 65 years with a clinical diagnosis of TMD associated with pain for at least three months and bruxism. All participants must provide informed consent prior to inclusion. Individuals with congenital malformations or cervical spine pathology, acute infectious or inflammatory disease, vestibular dysfunction, technical contraindications, recent manual therapy treatment (within one month), or recent use of analgesic, muscle relaxant, or anti-inflammatory medication (within eight hours) will be excluded.

The study aims to determine whether the application of active mandibular techniques combined with specific cervical motor control training results in superior improvements in function and pain compared to standard clinical management. Furthermore, the analysis will consider sex-related differences in baseline characteristics and treatment outcomes. Results from this trial may provide clinically relevant evidence to guide physiotherapeutic approaches for patients with TMD and bruxism, potentially improving therapeutic decision-making and long-term patient outcomes. The findings will be disseminated through publication in high-impact international journals and presentation at scientific conferences.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Clinical diagnosis of temporomandibular disorder and/or bruxism.
* Presence of pain and/or functional limitation.
* Ability to provide informed consent.
* Willingness to participate in the exercise program.

Exclusion Criteria:

* Previous surgery or major trauma to the cervical or maxillofacial area.
* Neurological disorders affecting motor control.
* Severe psychiatric disorders.
* Active inflammatory or rheumatologic conditions of the temporomandibular joint.
* Ongoing physiotherapeutic treatment targeting the studied region.
* Anti-inflammatory treatment 8 hours or less before the study.
* Pregnancy
* Inability to comply with the intervention protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT / UDP) | After 4-week intervention and 12 week follow up.
  The primary outcome will be the change in pressure pain threshold (PPT), also referred to as Umbral de Dolor a la Presión (UDP), measured in kg/cm² using a handheld pressure algometer at clinically relevant trigger points of the upper trapezius, masseter, external pterygoid, and digastric muscles. An increase in PPT indicates improved pain sensitivity. The objective is to determine whether the mandibular muscle energy technique combined with cranio-cervical control exercise leads to superior improvements compared to standard care and placebo suboccipital inhibition techniques

SECONDARY OUTCOMES:
Maximum Mouth Opening (MMO) | Baseline, after 4-week intervention, 12 week follow up.
  Maximum mouth opening will be measured in millimeters using a digital caliper or equivalent device. Measurements will be taken during active mandibular depression without pain-provocation, and repeated at baseline, after 4 weeks of treatment, and at follow-up. Improved range of mandibular motion is an indicator of enhanced temporomandibular functionality. Previous research cited in the protocol indicates that motor interventions directed at the cervical spine and mandibular musculature have been associated with increases in mouth opening capacity.
Pain Intensity | Baseline, after 4-week intervention and at 12 week follow up.
  Pain intensity will be quantified using a validated subjective scale such as Visual Analog Scale (VAS) or Numeric Pain Rating Scale. VAS is a simple, 1-dimensional measurement tool used to assess subjective experiences like pain, fatigue, or mood, typically a 10-centimeter line with descriptive anchors (e.g., "no pain" to "worst imaginable pain") at each end, where patients mark their current feeling, and clinicians measure the distance from the start to get a score (0-10 or 0-100). The NPRS is a simple 11-point scale (0-10) where patients rate their pain intensity, with 0 being "no pain" and 10 being the "worst pain imaginable", helping clinicians track pain levels and treatment effectiveness. Pain reduction is expected as a direct result of the active mandibular and cervical therapeutic exercises, which have previously demonstrated improvements in patients with temporomandibular disorders.
Craniocervical Postural Control | Baseline, after 4-week intervention and at 12 week follow up.
  Postural control of the craniocervical region will be assessed through standardized tests of cervical motor control and alignment (e.g., deep cervical flexor endurance test, joint repositioning accuracy, or similar). Baseline and post-intervention evaluations will determine whether targeting mandibular musculature in combination with cervical stabilization exercises contributes to improved neuromuscular coordination and postural balance. This is supported by previous studies showing multidirectional effects between cervical and mandibular systems.
Mandibular Range of Motion | Baseline, after 4-week intervention and at 12 week follow up.
  Mandibular movements will be assessed using a digital caliper, with measurements recorded in millimeters (mm). Movements evaluated will include maximum mouth opening and left and right lateral deviation. For each movement, two to three individual measurements will be obtained, and the mean value will be calculated for analysis. Measurements will be collected pre and post intervention, allowing for evaluation of changes in mandibular mobility.
Myofascial Trigger Point Sensitivity | Baseline, after 4-week intervention and at 12 week follow up.
  Pressure pain threshold (PPT) of myofascial trigger points in the main mandibular muscles will be measured using a pressure algometer. The algometer quantifies the pressure required to elicit pain at a specific muscular trigger point, expressed in kg/cm². Measurements will be obtained bilaterally, including both the left and right hemiface, and recorded pre and post intervention. Higher PPT values indicate lower sensitivity or pain at the trigger point, whereas lower values indicate higher sensitivity.
Cervical Motor Control | Baseline, after 4-week intervention and at 12 week follow up.
  Cervical motor control evaluates the range of motion in flexion, extension, and right and left cervical rotation. It will be evaluated by measuring movement deviations during a motor control task. Deviations from a visual target will be recorded in centimeters (cm). Larger deviations indicate poorer motor control, while smaller deviations indicate better accuracy and control. Measurements will be collected pre and post intervention.
Fear of Movement | Baseline, after 4-week intervention and at 12 week follow up.
  Fear of movement and pain-related avoidance behaviors will be assessed using the Tampa Scale for Kinesiophobia (TSK) and the Visual Analogue Scale (VAS):
  TSK: A 17-item questionnaire that evaluates fear of movement and re-injury. Scores range from 17 to 68, with higher scores indicating greater kinesiophobia and fear of movement.
  VAS: A 10-cm visual scale measuring perceived pain or fear associated with movement. Scores range from 0 (no fear/pain) to 10 (maximum fear/pain).
  Both scales will be used pre and post intervention, allowing assessment of changes in fear and pain perception over time.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Márquez Vera, PhD, Principal Investigator — Centro Asistencial Universitario de Salamanca (CAUSA); Jose Antonio Blanco Rueda, MD, PhD, Principal Investigator — Centro Asistencial Universitario de Salamanca (CAUSA)
Locations (1):
- Complejo Asistencial Universitario de Salamanca, Salamanca, Salamanca, Spain

REFERENCES:
- [Background] Mansilla-Ferragut P, Fernandez-de-Las Penas C, Alburquerque-Sendin F, Cleland JA, Bosca-Gandia JJ. Immediate effects of atlanto-occipital joint manipulation on active mouth opening and pressure pain sensitivity in women with mechanical neck pain. J Manipulative Physiol Ther. 2009 Feb;32(2):101-6. doi: 10.1016/j.jmpt.2008.12.003. PMID 19243721
- [Background] Mansilla Ferragut P, Boscá Gandía JJ. Efecto de la manipulación de la charnela occipito-atlo-axoidea en la apertura de la boca. Osteopatía Científica. 2008;3(2):45-51.
- [Background] Bretischwerdt C, Rivas-Cano L, Palomeque-del-Cerro L, Fernandez-de-las-Penas C, Alburquerque-Sendin F. Immediate effects of hamstring muscle stretching on pressure pain sensitivity and active mouth opening in healthy subjects. J Manipulative Physiol Ther. 2010 Jan;33(1):42-7. doi: 10.1016/j.jmpt.2009.11.009. PMID 20114099
- [Background] Whittingham W, Nilsson N. Active range of motion in the cervical spine increases after spinal manipulation (toggle recoil). J Manipulative Physiol Ther. 2001 Nov-Dec;24(9):552-5. doi: 10.1067/mmt.2001.118979. PMID 11753327
- [Background] Gross A, Miller J, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL; COG. Manipulation or mobilisation for neck pain: a Cochrane Review. Man Ther. 2010 Aug;15(4):315-33. doi: 10.1016/j.math.2010.04.002. Epub 2010 May 26. PMID 20510644
- [Background] 17. Fernandes Juca K, Claudio Suazo Galdames I. Posición Condilar en Apertura Oral Máxima. Una Evaluación con Imágenes de Resonancia Magnética. Int. J. Morphol. 2009; 27(3):867-71.
- [Background] Fey MF. [Diagnostic DNA probes]. Schweiz Med Wochenschr. 1990 May 19;120(20):731-7. German. PMID 2190309
- [Background] 15. Jiménez-Silva A, Peña-Durán C, Lee-Munoz X, Vergara-Núnez C, Tobar-Reyes J y Frugone-Zambra R. Patología temporomandibular asociada a masticación unilateral en adultos jóvenes. Rev Clin Periodoncia Implantol Rehabil Oral. 2016;9(2):125-31.
- [Background] Aparicio EQ, Quirante LB, Blanco CR, Sendin FA. Immediate effects of the suboccipital muscle inhibition technique in subjects with short hamstring syndrome. J Manipulative Physiol Ther. 2009 May;32(4):262-9. doi: 10.1016/j.jmpt.2009.03.006. PMID 19447262
- [Background] 12. Rodríguez Blanco C, Torres-Lagares D, Munuera Martínez PV, Oliva Pascual-Vaca A. Influencias de la relación maxilomandibular en el tratamiento postural mediante inhibición muscular. Osteopatía Científica. 2009;4(3):115-119
- [Background] 11. Gerez J, Figallo MA, Martínez PV, Rabadán M, Ortega MÁ, Vidal JA, Hernández MS. Short Term Application of the Muscular Inhibition Method of Strain/Counterstrain in the Treatment of Latent Myofascial Trigger Points of the Masticatory Musculature: A Randomized Controlled Trial. Clin Adv in Health Res. 2019; 1.1: 2-10.
- [Background] Armijo-Olivo S, Pitance L, Singh V, Neto F, Thie N, Michelotti A. Effectiveness of Manual Therapy and Therapeutic Exercise for Temporomandibular Disorders: Systematic Review and Meta-Analysis. Phys Ther. 2016 Jan;96(1):9-25. doi: 10.2522/ptj.20140548. Epub 2015 Aug 20. PMID 26294683
- [Background] Olivo SA, Fuentes J, Major PW, Warren S, Thie NM, Magee DJ. The association between neck disability and jaw disability. J Oral Rehabil. 2010 Sep;37(9):670-9. doi: 10.1111/j.1365-2842.2010.02098.x. Epub 2010 May 27. PMID 20524969
- [Background] Gencosmanoglu H, Unluer NO, Akin ME, Demir P, Aydin G. An investigation of biomechanics, muscle performance, and disability level of craniocervical region of individuals with temporomandibular disorder. Cranio. 2024 Mar;42(2):232-242. doi: 10.1080/08869634.2021.1938854. Epub 2021 Jun 15. PMID 34128775
- [Background] 7. Cocera Morata F, Rodríguez Blanco C. Relaciones entre la patología suboccipital y los trastornos temporomandibulares en el tratamiento osteopático. Osteopatía Científica. 2014;9(3):60-66.
- [Background] 6. Oliva Pascual-Vaca A, Rodríguez Blanco C. Sistema estomatognático, osteopatía y postura. Osteopatía Científica. 2008;3(2):88-90.
- [Background] 4. Hormiga Sánchez C, Bonet Collante M, Alodia Martínez C. Prevalencia de síntomas y signos de trastornos temporomandibulares en una población universitaria del área metropolitana de Bucamango, Santander. Umbral Científico, Bogotá Colombia. Junio de 2009: (14) 80-91.
- [Background] 2. Bermejo-Fenoll A. Desórdenes temporomandibulares. Madrid: Science Tools; 2008.
- [Background] 1. Rodríguez-Ozores Sánchez R. Mejorando la capacidad resolutiva. Patología de la Articulación Temporomandibular. Madrid, AMF, 2010: (6) 599-658.